CLINICAL TRIAL: NCT07106437
Title: Assessing Waste and Environmental Impact in Catheterization Laboratories: Results From the GREEN CATHeter Lab Study
Brief Title: GREEN CATHeter Lab Study
Acronym: GREEN-CATH
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: kt25Boeddinghaus2
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Waste, Medical; Waste, Procedural
Keywords: ecological footprint; Interventional cardiology procedures; environmental impact; CO₂ emissions; disposal costs; ReCiPe endpoint method; life cycle impact assessment

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Elective diagnostic coronary angiography: Elective diagnostic coronary angiography with or without simple PCI
  Interventions: Other: "Basel Model": Measure of total waste after completion of the procedure; Other: "Standard Model": Measure of total waste after completion of the procedure
- Complex percutaneous coronary interventions (PCI) procedures: Complex PCI procedures, including CTO, CHIP, or patients in cardiogenic shock requiring temporary mechanical circulatory support with an Impella device
  Interventions: Other: "Basel Model": Measure of total waste after completion of the procedure; Other: "Standard Model": Measure of total waste after completion of the procedure
- Structural heart intervention: transcatheter aortic valve implantation (TAVI): Structural heart intervention: TAVI
  Interventions: Other: "Basel Model": Measure of total waste after completion of the procedure; Other: "Standard Model": Measure of total waste after completion of the procedure
- Structural heart interventions: transcatheter edge-to-edge repair (TEER): Structural heart interventions: TEER of the mitral or tricuspid valves (MitraClip or TriClip systems)
  Interventions: Other: "Basel Model": Measure of total waste after completion of the procedure; Other: "Standard Model": Measure of total waste after completion of the procedure

INTERVENTIONS:
Other: "Basel Model": Measure of total waste after completion of the procedure — For each included case, the total waste generated will be measured in kilograms immediately after completion of the procedure and physically recorded by category in accordance with four predefined waste types: (i) paper and cardboard, (ii) regular waste (i.e., municipal solid waste or general trash), (iii) regulated medical waste (requiring specialized incineration including sharpsafe), and (iv) recyclable plastic
Other: "Standard Model": Measure of total waste after completion of the procedure — Simulation of a hypothetical but common practice in many hospitals, in which all waste generated during interventional procedures is disposed of as regulated medical waste, without separation.

SUMMARY:
This study involves the prospective quantification and classification of waste produced during interventional cardiology procedures. For each included case, the total waste generated will be measured in kilograms immediately after completion of the procedure. Waste will be physically sorted and recorded by category in accordance with four predefined waste types: (i) paper and cardboard, (ii) regular waste (i.e., municipal solid waste or general trash), (iii) regulated medical waste (requiring specialized incineration including sharpsafe), and (iv) recyclable plastic. Based on two models ("Basel Model" and "Standard Model"), the study will perform scenario-based calculations to compare the environmental and economic impact of both strategies.

DETAILED DESCRIPTION:
Interventional cardiology procedures generate substantial amounts of waste, not only medical waste but also large volumes of packaging materials such as paper, cardboard, and plastic. In many hospitals, all procedural waste, regardless of type, is disposed of as medical waste. This practice results in high disposal costs and increased environmental burden, as medical waste requires specialized, energy-intensive incineration and leads to considerable CO₂ emissions. At the University Hospital Basel, waste is systematically separated into categories, enabling structured evaluation of waste streams and environmental impact. Despite growing interest in sustainable healthcare, there is currently a lack of data on the quantity and composition of waste generated per specific procedure type in interventional cardiology. This creates an unmet need to quantify not only how much waste is produced but also to identify which components may be recyclable. this study is to quantify the total amount and type of waste generated during interventional cardiovascular procedures and to contextualize this waste in relation to the average daily waste production of both a Swiss resident and a hospital inpatient. By linking procedural waste generation to familiar population-based benchmarks, This study aims to provide a comprehensible measure of the environmental footprint of each procedure type. Waste will be recorded in kilograms and categorized into four predefined waste streams (paper/cardboard, regular municipal waste, regulated medical waste, and recyclable plastic). To ensure representative and comparable results, at least ten cases for each of the following procedure groups will be included: (i) elective coronary angiography with (ia) or without (ib) percutaneous coronary intervention (PCI), (ii) complex PCI procedures, such as chronic total occlusions (CTO), complex high-risk indicated procedures (CHIP), or interventions performed in patients with cardiogenic shock requiring mechanical support (e.g., Impella), and (iii) structural heart interventions, including TAVI and (iv) TEER of the mitral or tricuspid valves (MitraClip or TriClip).

To assess the broader ecological and financial implications of current waste management practices, two comparative disposal models will be applied. The first, referred to as the "Basel Model", reflects the current institutional practice at the University Hospital Basel, where procedural waste is systematically separated into the four aforementioned categories at the point of care. The second, the "Standard Model", simulates a hypothetical but common practice in many hospitals, in which all waste generated during interventional procedures is disposed of as regulated medical waste, without separation.Based on these two models, the study will perform scenario-based calculations to compare the environmental and economic impact of both strategies.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing the following interventional procedures:

  o Elective diagnostic coronary angiography
* with PCI
* without PCI

  * Complex percutaneous coronary interventions (CTO, CHIP, or patients with cardiogenic shock requiring Impella support)
  * Structural heart intervention: TAVI
  * Structural heart interventions: TEER of the mitral or tricuspid valve (MitraClip or TriClip)

Exclusion Criteria:

* No exclusion criteria, as no patient-specific data are collected and no modifications to clinical care are introduced

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study "population" includes the following interventional procedures on scheduled audit days: (i) elective diagnostic coronary angiography with or without simple PCI, (ii) complex PCI procedures, including CTO, CHIP, or patients in cardiogenic shock requiring temporary mechanical circulatory support with an Impella device, (iii) TAVI, and (iv) TEER of the mitral or tricuspid valves, such as with MitraClip or TriClip systems. A minimum of ten cases per procedure type will be targeted to ensure adequate comparisons. All patients undergoing the above-listed procedures during the defined measurement days are eligible for inclusion
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Total amount of waste (kilogram) generated per cardiac intervention- procedure type | one time assessment immediately after cardiac intervention
  The waste will be weighed using a certified, hospital-grade scale provided by the in-house hospital pharmacy (Beurer, Typ KS 59, max 20 kg).
Composition of waste (by waste category) generated per cardiac intervention- procedure type | one time assessment immediately after cardiac intervention
  Waste will be physically sorted and recorded by category in accordance with four predefined waste types: (i) paper and cardboard, (ii) regular waste (i.e., municipal solid waste or general trash), (iii) regulated medical waste (requiring specialized incineration including sharpsafe), and (iv) recyclable plastic.
Relation of waste output to the average daily waste production of a Swiss resident (in kilogram) | one time assessment immediately after cardiac intervention
  Relation of waste output generated per cardiac intervention- procedure type to the average daily waste production of a Swiss resident (in kilogram)
Relation of waste output to the average daily waste production of a typical inhospital patient (in kilogram) | one time assessment immediately after cardiac intervention
  Relation of waste output generated per cardiac intervention- procedure type to the average daily waste production of a typical inhospital patient (in kilogram)

SECONDARY OUTCOMES:
Comparison of environmental impact by CO₂ emissions | Postprocedural (one time assessment after cardiac intervention)
  Environmental impact (CO₂ emissions) assuming no waste separation ("Standard model") compared with the structured separation model used at the University Hospital Basel ("Basel model")
Comparison of environmental impact by disposal costs (in Swiss Francs) | Postprocedural (one time assessment after cardiac intervention)
  Environmental impact (disposal costs) assuming no waste separation ("Standard model") compared with the structured separation model used at the University Hospital Basel ("Basel model")
Ecological burden by ReCiPe score | Postprocedural (one time assessment after cardiac intervention)
  Calculation of the ecological burden using ReCiPe score to provide standardized environmental impact score per procedure type (DALY, PDF/m²/yr, $). These values allow for comparison across material types and disposal processes.

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Boeddinghaus, PD Dr. med., Principal Investigator — Department of Cardiology, University Heart Center Basel, University Hospital Basel
Locations (1):
- Department of Cardiology, University Heart Center Basel, University Hospital Basel, Basel, Switzerland